CLINICAL TRIAL: NCT06573892
Title: Development of a Panel of Microbiome Markers for Predicting CHF Outcomes
Brief Title: The Gut Microbiome in Chronic Heart Failure
Acronym: GMCHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazarbayev University (Other)
Responsible Party: Principal Investigator, Almagul Kushugulova, specialist, Nazarbayev University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BR21882152
Record Dates: First submitted 2024-08-01; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The patient sample will be divided into three main groups based on clinical phenotypes determined by echocardiographic examination:
  HF with preserved ejection fraction (EF) (EF > 50%) HF with mildly reduced EF (EF 49-40%) HF with reduced EF (EF < 40%)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic. Heart Failure (Active Comparator): The patient sample will be divided into three main groups based on clinical phenotypes determined by echocardiographic examination:
  HF with preserved ejection fraction (EF) (EF > 50%) HF with mildly reduced EF (EF 49-40%) HF with reduced EF (EF < 40%) 30 patients in each group
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Placebo
- Placebo. Heart Failure (Placebo Comparator): The patient sample will be divided into three main groups based on clinical phenotypes determined by echocardiographic examination:
  HF with preserved ejection fraction (EF) (EF > 50%) HF with mildly reduced EF (EF 49-40%) HF with reduced EF (EF < 40%) 30 patients in each group
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Patients will receive the product twice a day, a single dose of the product is packaged in sachets. The product can be hired in the form of a powder or diluted with a small amount of water. The general course is 90 days.
  Other Names: mare's milk
Dietary Supplement: Placebo — Patients will receive the product twice a day, a single dose of the product is packaged in sachets. The product can be hired in the form of a powder or diluted with a small amount of water. The general course is 90 days.
  Other Names: caw milk

SUMMARY:
there are numerous studies, most of which are predominantly associative in nature, investigating the association between the gut microbiota and various pathologies. However, to establish a causal relationship between microbiome composition and chronic heart failure (HF), clinical studies are needed, particularly using probiotics that can modify the composition and function of the gut microbiota. Examining their effects on HF can help understand which specific changes are associated with improvement or slowing the progression of the disease. The gut microbiome plays an important role in regulating the immune system and inflammatory processes. Investigating the impact of probiotics on these mechanisms may reveal their potential anti-inflammatory and immunomodulatory properties, which can be beneficial for controlling the inflammation characteristic of HF. Additionally, studying the interaction of probiotics with other medications, such as antihypertensive and diuretic agents, can be crucial for optimizing pharmacotherapy in HF patients. Confirming the role of the gut microbiota in the pathogenesis of HF and further developing probiotic therapy may lead to improved prognosis and treatment outcomes for HF patients. Overall, conducting a clinical study using probiotics in HF has the potential to expand our knowledge of the role of the gut microbiota in this disease and lay the groundwork for the development of new treatment strategies.

DETAILED DESCRIPTION:
The patient sample will be divided into three main groups based on clinical phenotypes determined by echocardiographic examination:

HF with preserved ejection fraction (EF) (EF > 50%) HF with mildly reduced EF (EF 49-40%) HF with reduced EF (EF < 40%) From each subgroup, 60 patients will be randomly selected to participate in a double-blind, randomized, placebo-controlled trial of probiotic therapy.

The control group will consist of individuals selected from outpatient clinics in the city of Astana, matched by gender and age, who are healthy in terms of cardiovascular and other systemic pathologies, not in an acute phase of any illness, willing to participate in the study, and have signed informed consent.

For each patient, a medical history will be collected, a physical examination will be performed to assess their clinical condition, the severity of heart failure symptoms will be evaluated using a severity scale (ANA/ACC), functional classes will be determined according to NYHA (6-minute walk test), echocardiographic examination will be conducted, and if indicated, electrocardiogram (ECG) monitoring using a Holter monitor will be performed. The physical examination will include lung auscultation, cardiac auscultation, assessment of peripheral edema, assessment of jugular venous pulse height, body weight, height, and height at the age of 20. Further investigations will be guided by symptoms. Echocardiographic examination will be performed using a diagnostic ultrasound device, Philips Ultrasound Inc., CX50. The 12-lead ECG will be recorded in the supine position. ECG intervals (PR, QRS, QT, QTc), heart rate, and any abnormalities (rhythm anomalies, AV block, pathological Q waves, bundle branch block, repolarization disturbances) will be recorded for each subject.

Clinical and laboratory parameters:

The following analyses will be performed:

* Complete blood count with differential leukocyte count
* Total/direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), lactate dehydrogenase (LDH)
* Total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglycerides
* Serum glucose, glycosylated hemoglobin (HbA1c)
* Blood electrolytes (sodium, potassium, chloride), creatinine, blood urea nitrogen (BUN), uric acid
* Glutamic-oxaloacetic transaminase, glutamic-pyruvic transaminase, gamma-glutamyl transferase (GGT)
* Creatine phosphokinase, troponin I
* Thyroid-stimulating hormone (TSH), triiodothyronine (T3), thyroxine (T4)

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Residing in the city of Astana and surrounding regions (Akmola region)
* Diagnosis of heart failure according to internationally recognized guidelines and classified as Class I-IV by NYHA (New York Heart Association) or Stage A-C according to ACC/AHA (American College of Cardiology/American Heart Association) classification
* Clinically stable condition and optimized medication therapy for heart failure for at least 4 weeks in accordance with current recommendations
* Willingness to participate in the study

Exclusion Criteria:

* • Age under 18 years

  * Refusal to undergo diagnostic procedures specified in the study protocol
  * Terminal stage of heart failure (Stage D according to ACC/AHA classification)
  * Coronary or peripheral revascularization procedures, valvular procedures, or any major surgical procedure within 3 months prior to study enrollment
  * Use of antibiotics, cytostatic therapy, or pro- or prebiotics within 1 month prior to the baseline visit
  * Presence of oncological and autoimmune diseases (connective tissue diseases, gastrointestinal disorders, skin disorders, etc.)
  * Acute illness or active infection
  * Individual intolerance to the administered nutrients (probiotics)
  * Presence of other anatomical or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, may limit the subject's ability to participate in the clinical study, comply with the requirements of subsequent follow-up, or affect the scientific validity of the clinical study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | 90 days
  Changes in gut microbiota composition [Timepoints: baseline, after 3 months of probiotic intake]

SECONDARY OUTCOMES:
Frequency of hospitalizations | 2 years
  Frequency of hospitalizations and cardiovascular mortality [Timepoints: baseline, after 3 months of probiotic intake]

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Issilbayeva A, Sergazy S, Zhashkeyev A, Gulyayev A, Kozhakhmetov S, Shulgau Z, Nurgaziyev M, Nurgaziyeva A, Zhetkenev S, Mukhanbetzhanov N, Jarmukhanov Z, Mukhanbetzhanova Z, Vinogradova E, Zhumadilov Z, Kushugulova A, Aljofan M. Polyphenol-mediated microbiome modulation in STEMI patients: a pilot study. Front Med (Lausanne). 2025 May 21;12:1522373. doi: 10.3389/fmed.2025.1522373. eCollection 2025. PMID 40470050